CLINICAL TRIAL: NCT02299882
Title: Surgical Infection Rates With Adjunct Vancomycin Compared to Standard Peri-Operative IV Antibiotics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corewell Health West (Other)
Responsible Party: Principal Investigator, Jason A Squires, DO, Physician, Corewell Health West
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2012-166
Record Dates: First submitted 2013-02-20; First posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2013-02

CONDITIONS: Lumbar Pain
Keywords: Posterior spine surgery; infection; vancomycin; surgical wound infection
MeSH Terms: conditions — Low Back Pain; Infections; Surgical Wound Infection | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vancomycin (Experimental): Patient will receive Vancomycin powder to the incision just before skin closure
  Interventions: Drug: Vancomycin
- no vancomycin (No Intervention): Patient will be randomized to either vancomycin powder or no vancomycin powder. This arm the patient will not have the powder placed in the incision before skin closure.

INTERVENTIONS:
Drug: Vancomycin — Patient will be randomized to either vancomycin or no vancomycin. This treatment will take place prior to the closure of the incision from back surgery.
  Arms: Vancomycin

SUMMARY:
Determine the effect of Vancomycin Powder added to the surgical wound at closure on surgical infection rates.

DETAILED DESCRIPTION:
Study will be blinded and randomized 1:1 to either Vancomycin Powder at closure or no vancomycin powder at closure.

ELIGIBILITY:
Inclusion Criteria:

* All adult, 18 years or greater undergoing posterior approach spinal surgery

Exclusion Criteria:

* Prisoner, pregnant women, patient under the age of 18, those of diminished decision making capacity.
* patients with known reaction to Vancomycin.
* patients having surgery specifically for spine infection
* patients having ADCF or ALIF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-08 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Surgical wound infection rate, both deep and superficial infections | 12 weeks post surgery

SECONDARY OUTCOMES:
Post-operative rate of MRSA infections. | 12 weeks post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jason Squires, DO, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health Hospitals, Grand Rapids, Michigan, United States